CLINICAL TRIAL: NCT00031863
Title: Phase III, Randomized, Double Blind, Placebo Controlled Study of Rofecoxib in Colorectal Cancer Patients Following Adjuvant Chemotherapy
Brief Title: Rofecoxib After Surgery in Treating Patients With Stage II or Stage III Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cancer Research Campaign Clinical Trials Centre (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: CRC-TU-VICTOR; CDR0000069235 (Registry Identifier: PDQ (Physician Data Query)); EU-20054; CRC-TU-COX2; ISRCTN98278138; NCCTG-N004B
Record Dates: First submitted 2002-03-08; First posted 2003-01-27 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2002-06

CONDITIONS: Colorectal Cancer
Keywords: stage II colon cancer; stage III colon cancer; stage II rectal cancer; stage III rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — rofecoxib; Chemotherapy, Adjuvant

INTERVENTIONS:
Drug: rofecoxib
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Rofecoxib may stop the growth of cancer by stopping blood flow to the tumor and killing tumor cells that remain after surgery. It is not yet known if rofecoxib is effective in treating colorectal cancer.

PURPOSE: Randomized phase III trial to determine the effectiveness of giving rofecoxib after surgery in treating patients who have stage II or stage III colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall survival of patients with previously resected stage II or III colorectal cancer treated with rofecoxib vs placebo administered for at least 2 years vs 5 years.
* Compare the relapse-free survival of patients treated with these regimens.

OUTLINE: This is a randomized, placebo-controlled, double-blind, multicenter study. Patients are stratified according to participating center, site of disease (colon vs rectum), disease stage (II vs III), age, adjuvant chemotherapy (yes vs no), and type of chemotherapy regimen (1 vs 2 vs 3 vs 4 vs 5). Within 3 months of surgical resection alone or completion of adjuvant radiotherapy and/or chemotherapy after surgical resection, patients are randomized to one of four treatment arms.

* Arm I: Patients receive oral rofecoxib once daily for 2 years.
* Arm II: Patients receive oral rofecoxib once daily for 5 years.
* Arm III: Patients receive oral placebo once daily for 2 years.
* Arm IV: Patients receive oral placebo once daily for 5 years. Treatment continues in all arms in the absence of disease recurrence or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 7,000 patients (1,750 per treatment arm) will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed colorectal carcinoma

  * Stage II (T3-4, N0, M0) or stage III (any T, N1-2, M0) disease
* Completely resected primary tumor without gross or microscopic evidence of residual disease
* Must have received potentially curative therapy within the past 12 weeks, including any of the following:

  * Surgery alone
  * Surgery plus radiotherapy and/or chemotherapy

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* WHO 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST/ALT no greater than 1.5 times ULN

Renal:

* Creatinine clearance greater than 30 mL/min

Cardiovascular:

* No severe congestive heart failure

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No active peptic ulcer or gastrointestinal bleeding within the past year
* No inflammatory bowel disease
* No known sensitivity to rofecoxib
* No prior adverse reaction to non-steroidal anti-inflammatory drugs (NSAIDs) (e.g., asthma, acute rhinitis, nasal polyps, angioneurotic edema, or urticaria)
* No other malignancy within the past 10 years except adequately treated carcinoma in situ of the cervix or basal cell or squamous cell skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics

Surgery:

* See Disease Characteristics

Other:

* No concurrent long-term NSAIDs except low-dose aspirin (no more than 80 mg/day) for cardio-prophylaxis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-02; Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J. Kerr, MD, FRCP, DSc, Study Chair — Oxford University Hospitals NHS Trust
Locations (1):
- Radcliffe Infirmary NHS Trust, Oxford, England, United Kingdom

REFERENCES:
- [Result] Midgley RS, McConkey CC, Johnstone EC, Dunn JA, Smith JL, Grumett SA, Julier P, Iveson C, Yanagisawa Y, Warren B, Langman MJ, Kerr DJ. Phase III randomized trial assessing rofecoxib in the adjuvant setting of colorectal cancer: final results of the VICTOR trial. J Clin Oncol. 2010 Oct 20;28(30):4575-80. doi: 10.1200/JCO.2010.29.6244. Epub 2010 Sep 13. PMID 20837956
- [Result] Kerr DJ, Dunn JA, Langman MJ, Smith JL, Midgley RS, Stanley A, Stokes JC, Julier P, Iveson C, Duvvuri R, McConkey CC; VICTOR Trial Group. Rofecoxib and cardiovascular adverse events in adjuvant treatment of colorectal cancer. N Engl J Med. 2007 Jul 26;357(4):360-9. doi: 10.1056/NEJMoa071841. PMID 17652651